CLINICAL TRIAL: NCT01015404
Title: A Study to Assess the Safety of Using Fibroblast Growth Factor-2 With Periodontal Surgery in Japan (Phase 3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaken Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCB-1D-04
Record Dates: First submitted 2009-11-16; First posted 2009-11-18 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Periodontitis
Keywords: Trafermin; Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — trafermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental H (Experimental): high volume (0.6mL、0.3% Trafermin)
  Interventions: Drug: Trafermin
- Experimental L (Experimental): low volume (0.2mL、0.3% Trafermin)
  Interventions: Drug: Trafermin

INTERVENTIONS:
Drug: Trafermin — Administered to the bone defect during flap operation
  Other Names: KCB-1D

SUMMARY:
This study aims to investigate the safety in using Trafermin (recombinant human basic fibroblast growth factor) with periodontal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Vertical intrabony defect from radiographs at baseline
* Age of 20 years or older

Exclusion Criteria:

* Using an investigational drug within the past 24 months
* Coexisting malignant tumour or history of the same
* Coexisting diabetes (HbA1C 6.5% or more)
* Taking bisphosphonates
* Coexisting gingival overgrowth or history of the same

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
serum Trafermin level | within 4 weeks

SECONDARY OUTCOMES:
occurrence and level of adverse reaction | within 4 weeks
serum anti-Trafermin antibody level | within 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chikara Ieda, Study Director — Kaken Pharmaceutical Co., Ltd.
Locations (6):
- Japan (6):
  - Kaken Investigational Site 5, Chiyoda-ku
  - Kaken Investigational Site 2, Matsudo
  - Kaken Investigational Site 3, Ōta-ku
  - Kaken Investigational Site 1, Sapporo
  - Kaken Investigational Site 4, Shinjuku-ku
  - Kaken Investigational Site 6, Suita

REFERENCES:
- [Result] Kitamura M, Nakashima K, Kowashi Y, Fujii T, Shimauchi H, Sasano T, Furuuchi T, Fukuda M, Noguchi T, Shibutani T, Iwayama Y, Takashiba S, Kurihara H, Ninomiya M, Kido J, Nagata T, Hamachi T, Maeda K, Hara Y, Izumi Y, Hirofuji T, Imai E, Omae M, Watanuki M, Murakami S. Periodontal tissue regeneration using fibroblast growth factor-2: randomized controlled phase II clinical trial. PLoS One. 2008 Jul 2;3(7):e2611. doi: 10.1371/journal.pone.0002611. PMID 18596969